CLINICAL TRIAL: NCT05539482
Title: A Multicenter, Cluster-Randomized, Active-Controlled, Single-Blind Trial of Community-Based Health Education Programs for the Early Detection of, and Vaccination Against, COVID-19 and the Adoption of Self-Protective Measures of Hong Kong Residents
Brief Title: Community-Based Health Education Programs for the Early Detection of, and Vaccination Against, COVID-19 and the Adoption of Self-Protective Measures of Hong Kong Residents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, XIE Yao Jie Grace, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P0039048; COVID1903006-A (Other Grant/Funding Number: HMRF)
Record Dates: First submitted 2022-09-04; First posted 2022-09-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: CBPR; health education; vaccination rate; early-testing; self-protection; Hong Kong residents
MeSH Terms: conditions — COVID-19; Health Education

STUDY DESIGN:
Intervention Model Description: The participants recruited by one collaborator will be considered as one cluster. A research assistant will randomly assign the clusters from the NGOs, Schools, and Companies to either the intervention group or the active control group, respectively. After allocation, there will be four clusters in both the intervention and control groups from the NGOs, schools and companies, respectively. This will result in 3 × 4 = 12 clusters for each group (intervention/control). A active control group will be used instead of a standard control group to help motivate the collaborators to implement the program and to avoid a high participant dropout rate.
Who Masked: Participant
Masking Description: All the participants will be blind to the allocation. Participants in the intervention group will receive intervention based on core package, while participants in the control will receive health information which are collected and provided by collaborators. The collaborator also will be told to avoid discussing allocation with the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community-Based Health Education Group (Experimental): The collaborators will design the Community-based education approach (based on the core intervention package). Collaborators will be required to submit a brief standardized proposal to the academic investigators for review and approval, to ensure that all intervention programs have the same core intervention content and can be implemented appropriately. Collaborators will be able to use any reasonable strategies, such as social media platforms, information technology, posters, leaflets, and videos, to implement the programs . The use of incentives will be encouraged to improve participation. Each programs will last for 3 months. A booster session will be conducted at the mid of the intervention.
  Interventions: Behavioral: Community-based Health Education based on core intervention package
- Health Information Sharing Group (Active Comparator): The collaborators will design the community-based education approach and deliver health information to the participants. Researchers will provide some information, while collaborators need to self-collect the rest. Collaborators also need to submit a proposal to ensure the feasibility of intervention programs and the accuracy of health information. Collaborators can use any reasonable strategies to implement the programs . The use of incentives will be encouraged to improve participation. Each programs will last for 3 months. A booster session will be conducted at the mid of the intervention.
  Interventions: Behavioral: Health Information Sharing Group

INTERVENTIONS:
Behavioral: Community-based Health Education based on core intervention package — Community-based Health Education will potentially include the following three components:
  1. A manual of emergency preparedness and self-protection against COVID-19 infection. The main content will include hand washing, mask wearing and social distancing guidelines.
  2. Early testing. Participants will be trained on how to recognize the early symptoms of COVID-19 and appropriate practice to take in a response, and they will be provided with testing resources.
  3. Knowledge of vaccines and their benefits and resources for vaccination.
  Collaborators should design and implement health programs based on the core intervention package.
  Arms: Community-Based Health Education Group
Behavioral: Health Information Sharing Group — Collaborators are encouraged to collect and share health information to the participants. Shared information should be previewed by researchers.
  Arms: Health Information Sharing Group

SUMMARY:
This study evaluates the community-based health education program in improving early testing for COVID-19, increasing vaccination acceptability and enhancing emergency preparedness and self-protection measures against COVID-19 in HK. We established a partnership with several local community stakeholders and they will be responsible for recruiting participants and implementing educational programs. Half of the community collaborators will receive the core intervention package, and use it as education material. The other half will be encouraged to self-collect and send health information to the participants.

DETAILED DESCRIPTION:
This health education program is based on a Community-based Participants Research (CBPR) approach, which is a partnership approach that equitably involves community members and researchers in all aspects of the research process. Given the different cultural, professional or living background of Hong Kong residents, we think this simple, flexible and sustainable approach will effectively mitigate the COVID-19 risk in HK society,

An academic-community collaboration platform with several nongovernmental organizations (NGOs), companies and schools will be established before this study. They will work together to recruit participants, design and implement a series of educational programs aimed at controlling the spread of COVID-19 in the community.

ELIGIBILITY:
For participants recruited by NGOs and companies, the Inclusion Criteria will be:

* HK resident aged 18 years or above;
* Agreement to participate in the study and provide written informed consent.

The Exclusion Criteria will be:

* Cognitive impairment that inhibits communication with the investigators;
* Inability or unwillingness to provide written informed consent.

For participants recruited by schools, the Inclusion Criteria will be:

* HK students aged 12 to 18 years and their parents.

The Exclusion Criteria will be:

* Cannot provide written informed consent (or assent for the younger students).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Vaccination rates | 3 months
  The number of participants who received a new dose of COVID-19 vaccine over the total number of participants.

SECONDARY OUTCOMES:
The knowledge towards COVID-19 vaccine | 3 months
  The knowledge towards COVID-19 vaccine will be measured by 15 items in the self-administered questionnaire. All the items are binary- choice Items (1=Ture, 2= False). The total score ranged from 15 to 30 and a higher score indicates poorer knowledge towards COVID-19 vaccine.
The hesitancy towards COVID-19 vaccine | 3 months
  The hesitancy towards COVID-19 vaccine will be measured by Chinese version of adult Vaccine Hesitancy Scale (aVAS), which includes 10 items of 5-point Likert scale, ranging from least hesitant (1) to most hesitant (5). In total 3 of aVAS are negatively worded and 7 are positively worded. The total score of aVAS is 50 with a score higher than 25 indicated high vaccine hesitancy.
Perceived confidence of COVID-19 vaccine | 3 months
  The confidence of COVID-19 vaccine will be measured by 11 items with 5-point Likert scale with "strongly disagree", "disagree", "neither agree nor disagree", "agree" and "strongly agree". The total score ranges from 11 to 55 with higher score indicating higher confidence of COVID-19 vaccine..
Perceived barriers of receiving COVID-19 vaccine | 3 months
  The perceived barriers of COVID-19 vaccine will be measured by 4 items with 5-point Likert scale with "strongly disagree", "disagree", "neither agree nor disagree", "agree" and "strongly agree". The total score ranges from 4 to 20 with higher score indicating higher perceived barriers of COVID-19 vaccine..
The amount of early testing | 3 months
  The amount of early testing will be measured by self-reported number of early-testing with rapid antigen testing (RAT) in a month.
The levels of acceptability for early testing | 3 months
  The levels of acceptability for early testing will be measured by 3 items with 5-point Likert scale with "strongly disagree", "disagree", "neither agree nor disagree", "agree" and "strongly agree". The total score ranges from 3 to 15 with higher score indicating higher acceptability of early testing.
The frequency of washing hands with soap or hand sanitizer | 3 months
  The amount of early testing will be measured by self-reported number of hand-washing behaviors with soap or hand sanitizer per day in the past week.
The frequency of washing hands with alcohol-based hand rub | 3 months
  The amount of early testing will be measured by self-reported number of hand-washing behaviors with alcohol-based hand rub per day in the past week.
The knowledge of proper self-protection | 3 months
  The knowledge of proper self-protection correctly will be measured 13 items in the self-administered questionnaire. All the items are binary- choice Items (1=Ture, 2= False). The total score ranged from 13 to 26 and a higher score indicates poorer knowledge of self-protection.
Stress status | 3 months
  The Perceived Stress Scale (PSS-4) will be used to measure the stress level.
Anxiety status | 3 months
  Generalized Anxiety Disorder (GAD-2) will be used to measure the level of anxiety.
Depression status | 3 months
  The Patient Health Questionnaire-2 (PHQ-2) will be used to measure the depression status.
Participants' satisfactory level | 3 months
  The participants' satisfactory level will be measured by asking the degree of satisfaction (1-10) in terms of vaccination, early-testing and self-protection.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Jie Xie, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Hong Kong

REFERENCES:
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249